CLINICAL TRIAL: NCT06434311
Title: Test-Retest Reliability and Concurrent Validity of the 3 Meter Backward Walk Test in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MarmaraU- AYDOĞDU-SÜZÜK001
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Knee Osteoarthritis: Patients who who have knee osteoarthritis categorized as 1 - 4 according to Kellgren - Lawrence
  Interventions: Diagnostic Test: 3 meter Backward Test

INTERVENTIONS:
Diagnostic Test: 3 meter Backward Test — evaluation

SUMMARY:
Osteoarthritis of the knee is a common joint disease that causes loss of balance and proprioception. Changes in the knee joint such as mechanoreceptor loss, muscle strength imbalance, muscle weakness, capsular hypertrophy, subchondral edema, and increased loss of balance and proprioception lead to an increased risk of falls. In the literature, knee osteoarthritis is repeatedly mentioned as an independent risk factor for falls, and knee osteoarthritis is associated with recurrent falls.

There are many performance-based clinical measurement tests that assess fall risk in knee osteoarthritis. Some of these tests include the timed up and walk test, the five-step sit-to-stand test, and the one-leg stand test. These tests cannot evaluate backward walking. Backward walking requires more neuromuscular control and proprioception than forward walking. The 3-meter backward walk test is a performance-based test that assesses backward walking, balance, proprioception, and neuromuscular control. The participant is asked to walk 3 meters backwards on a flat surface at the highest speed at which they feel comfortable without running. It is administered by recording the time elapsed.

The validity and reliability of the 3-meter walk back test have been previously investigated in many patient populations and healthy individuals. However, to our knowledge, there is no research on the reliability and validity of a 3-meter walk back test in knee osteoarthritis. Clinical measurement tests should be valid and reliable in the patient population to which they are applied.

The aim of this study was to examine the test-retest reliability and concurrent validity of the 3-meter backward walk test in participants with knee osteoarthritis. In addition, we aim to compare the 3-meter backward walk test scores of individuals with and without knee osteoarthritis and to examine the change in 3-meter backward walk test scores with the change in disease severity.

The data collection tools to be used in the study are the 3-meter walk back test, the timed get up and walk test, the Knee Injuries and Osteoarthritis Outcome Score, the Frail Scale, the Modified Falls Efficacy Scale, and fall history. All of these measures will be taken at the initial assessment, and the 3-meter walk back test will be repeated after 3-7 days.

We hope that our study will help physiotherapists working in this field in the clinical decision-making process by providing a valid and reliable performance test for the assessment of fall risk.

ELIGIBILITY:
Inclusion Criteria:

* To have been diagnosed with osteoarthritis by a specialist physician according to the clinical and radiological criteria of the American College of Rheumatology.
* Be between 40 and 75 years of age.
* Being in grade 1-4 according to Kellgren-Lawrence staging.
* To participate in the study voluntarily

Exclusion Criteria:

* Having undergone surgery involving the lower extremity
* Having prosthesis or orthosis in the lower extremity
* Other neurological and cardiopulmonary diseases that may affect walking and balance Having undergone surgery or invasive treatment in the last 6 months
* Body mass index above 45
* Having severe heart disease that prevents exercise
* Having pain originating from L3 - S1

Ages: 39 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have diagnosed as knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
3 meter Backward Test | At the baseline
  It is a performance-based test developed by Carter et al. A 3 meter long strip is drawn on the ground. It assesses fall risk, balance, neuromuscular control. Participants are expected to walk backwards for 3 meters as fast as possible. The time until the participant completes the walk is recorded. A lower score indicates higher performance (Carter et al., 2019).
3 meter Backward Test | One week later
  It is a performance-based test developed by Carter et al. A 3 meter long strip is drawn on the ground. It assesses fall risk, balance, neuromuscular control. Participants are expected to walk backwards for 3 meters as fast as possible. The time until the participant completes the walk is recorded. A lower score indicates higher performance (Carter et al., 2019).

SECONDARY OUTCOMES:
Timed Up Go Test | At the baseline
  The timed up and go test was developed in 1991 as a modified version of the get up and go test (Barry et al., 2014). The participant is asked to sit on a chair approximately 46 cm tall. Then, the participant gets up from the chair, walks 3 meters, walks the same distance back, and sits on the chair. The elapsed time is recorded (Barry et al., 2014; Ortega-Bastidas et al., 2023). A shorter time means a better score. The participant's failure to complete the test in less than 12 seconds indicates a high risk of falling (Nightingale et al., 2019).
Frail Scale | At the baseline
  It is a scale used to evaluate frailty in the elderly. The scale, consisting of 5 items, questions resistance, fatigue, ambulation, illness, and weight loss. Each question takes one of the values 0 or 1, with a total value of 0, indicating that the person is not frail. Values ranging from 1 to 2 are called pre-frail, and values above 2 are called fragile. In the disease questioning, the participant is asked how many of the 11 diseases he has. Having more than 5 diseases indicates a score of 1. The lowest score that can be obtained is zero, while the highest score is 5 (HYMABACCUS et al., 2023; Morley et al., 2012). Turkish validity and reliability study by Hymabaccus et al. Made by. Its reliability and validity have been reported as excellent, and the intraclass consistency coefficient varies between 0.68 and 0.82. (HYMABACCUS et al., 2023).
Knee injury and Osteoarthritis Outcome Score (KOOS) | At the Baseline
  It has been translated into more than fifty languages. The commonly used knee injury and osteoarthritis outcome score consists of 5 subcategories. It is a 5-point Likert type scale consisting of 42 questions. A score ranging from 0 to 4 is given for each question. The total score for each subcategory is one hundred. While 0 indicates serious knee problems, 100 indicates no knee problems (Roos, 2023). Turkish validity and reliability were determined by Paker et al. It was conducted in 2007 and reported moderate validity and reliability (Paker et al., 2007). Internal consistency was calculated with Cronbach's alpha and was reported as 0.66 - 0.95 (Paker et al., 2007).
Modified Falls Efficacy Scale | At the Baseline
  It evaluates the individual's self-confidence regarding the fall. It is an expanded version of the falls effectiveness scale. It consists of 14 items. It evaluates a person's self-confidence during various daily activities. Each item is given a value ranging from 0-10. While 0 represents unsafe, the number 10 is considered completely safe. The highest score that can be obtained is 140 and the lowest score is 0 (Soh et al., 2021). Turkish validity and reliability study by Korkmaz et al. Made by. The intra-class consistency coefficient was reported as 0.978 (Korkmaz et al., 2019).

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided